CLINICAL TRIAL: NCT00588172
Title: Genetic Variation in OCT1 and Response to Metformin
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Adrian Vella MD, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 07-004310; OCT1 and metformin
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Type 2 Diabetes
Keywords: Metformin; Type 2 diabetes; Oct1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Neurofibromatosis, Type 3, mixed central and peripheral | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Sham Comparator): Individuals with no nsSNPs or mutations known to alter oct1 function
  Interventions: Drug: Metformin
- 2 (Active Comparator): Individuals with nsSNPs or mutations known to alter oct1 function
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 1000mg bid for 1 week

SUMMARY:
Type 2 diabetes its microvascular and macrovascular complications have become a major global health problem. Metformin is often used as first-line therapy for this disorder given that it is cheap, may cause weight loss and does not have significant side-effects in healthy patients. On the other hand, as many as one third of all patients with type 2 diabetes initially treated with metformin never achieve a meaningful response to this intervention. Recently, genetic variation in the organic cation transporter 1 (Oct1) gene which encodes a protein, OCT1, mediating metformin uptake by the liver, its primary site of action, has been shown alter metformin action. In Oct1-deficient mice the glucose-lowering effects of metformin are completely abolished. Moreover a polymorphism with a 20% minor allele frequency in Caucasians also alters the effect of metformin on glucose tolerance (the net result of glucose uptake and glucose release) after ingestion of 75g of glucose. However, it is unknown if this polymorphism affects suppression of endogenous glucose production or stimulation of peripheral glucose uptake by metformin, or both, and to what degree. We propose to utilize established methodology to measure glucose turnover in response to a mixed meal to determine how common genetic variation in OCT1 alters response to metformin in healthy volunteers. This will clarify the effect of these variants on response to metformin in humans. The knowledge gained from this study will help to design future studies examining the role of OCT1 genotype in determining initial therapy for type 2 diabetes.

ELIGIBILITY:
Inclusion criteria: -

1. Heterozygous or homozygous for the nsSNPs R61C, G401S, 420Del, G465R, G174S (see supplementary info (3)) or without any nsSNPs that could potentially alter gene function.
2. Age 18 - 40.
3. Willingness to participate in this study.

Exclusion criteria: -

1. Fasting glucose > 100mg/dL on one occasion.
2. Use of medication other than stable thyroid hormone replacement or oral contraception.
3. Subjects must not be pregnant or < 6 months postpartum at the time of study.
4. Prior abdominal surgery other than hysterectomy, appendectomy or tubal ligation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Change in glucose area under the curve after a mixed meal in response to metformin | before and after 1 week of metformin

SECONDARY OUTCOMES:
Change in glucose disappearance and suppression of endogenous glucose production in response to metformin | before and after 1 week of metformin therapy

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic